CLINICAL TRIAL: NCT03670979
Title: A Novel Approach of Periodontal Osseous Wall Piezosplitting and EDTA Root Surface Etching in Management of Localized Intrabony Defects With Wide Angulation. Controlled Clinical Trial
Brief Title: Periodontal Osseous Wall Piezosplitting and EDTA Root Surface Etching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, mahmoud eldestawy, lecturer, periodontology department, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 839/2757
Record Dates: First submitted 2018-08-01; First posted 2018-09-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bone swaging alone (Experimental): xenograft alone
  Interventions: Procedure: bone swaging
- bone swaging plus EDTA (Experimental): bone swaging with EDTA
  Interventions: Procedure: bone swaging

INTERVENTIONS:
Procedure: bone swaging — osseous wall pedicle was placed to treat the infrabony defect by autogrnous bone

SUMMARY:
This study was designed to investigate the use of minimally invasive Piezo knife to harvest vascularized interceptal bone pedicle in treating intrabony defects.

DETAILED DESCRIPTION:
Sixteen non-smoking patients with severe chronic periodontitis participated in this prospective, randomized clinical study. Patients were randomly assigned into one of a 2 groups (8 patients each): bone substitute grafting of the intrabony defect, control group (Gr1), intrabony defect osseous wall swaging (OWS) combined xenograft (Gr2). In both groups root surfaces where treated with a neutral 24% EDTA gel and saline irrigation. Clinical and radiographic measurements were reassessed at 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. good compliance with plaque control instructions following initial therapy
2. teeth involved were all vital with no mobility ;
3. each subject contributed a single predominately 2 or 3-wall intrabony interproximal defect around premolar or molar teeth without furcation involvement;

Exclusion Criteria:

1. no systemic diseases which could influence the outcome of therapy;
2. absence of periodontal treatment during the previous year.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Radiographic evaluation | 3 months
  removing the defect as seen in radiograph defect filling with bone swaging with edta and bone substitute

SECONDARY OUTCOMES:
Clinical pocket depth | 3month
  By periodontal prob to measure the clinical parameter

CONTACTS AND LOCATIONS:
Overall Officials: ahmed y gamal, professor, Study Director — Ain Shams University

IPD SHARING:
Plan to Share IPD: Undecided
institutional review board, egypt